CLINICAL TRIAL: NCT05060991
Title: Impact of Immunosuppression Adjustment on the Immune Response to SARS-CoV-2 mRNA Vaccination in Kidney Transplant Recipients (ADIVKT)
Brief Title: Impact of Immunosuppression Adjustment on COVID-19 Vaccination Response in Kidney Transplant Recipients
Acronym: ADIVKT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: CareDx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1801321
Record Dates: First submitted 2021-09-24; First posted 2021-09-29 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Immunosuppression; Vaccine Response Impaired
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Prospective randomized open-labeled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Immunosuppression reduction (Experimental): Reduction of immunosuppression before and after administration of a third dose of SARS-CoV-2 mRNA vaccine
  Interventions: Drug: Reduction in antimetabolite immunosuppression
- Standard of care (No Intervention): No change to immunosuppression before or after receipt of a third dose of SARS-Co-2 mRNA vaccine

INTERVENTIONS:
Drug: Reduction in antimetabolite immunosuppression — Reduction in dose in mycophenolate mofetil/mycophenolic acid (MMF) or azathioprine before and after receiving 3rd dose vaccination
  Arms: Immunosuppression reduction

SUMMARY:
Immunocompromised individuals, such as solid organ transplant (SOT) recipients are at high risk of COVID-19 associated complications and mortality. Retrospective studies so far have shown that a majority of SOT recipients did not develop appreciable anti-spike antibody response after a first, second, or even third dose of mRNA vaccine. Treatment with antimetabolites was associated with poor vaccine response. The goal of this study is 1) examine whether transient immunosuppression reduction improves the immune response to a third dose of SARS-CoV-2 mRNA vaccine in kidney transplant recipients and 2) to assess the safety of immunosuppression reduction before and after third dose SARS-CoV-2 mRNA vaccination.

DETAILED DESCRIPTION:
This is a prospective, randomized open-labeled study of kidney transplant recipients who have previously received two doses of mRNA COVID-19 vaccine (either BNT162b2, Pfizer-BioNTech or mRNA-1273, Moderna) and who are eligible to receive a 3rd dose of mRNA vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* First or repeat kidney transplant recipient
* Negative or low positive antibody titer on SARS-CoV-2 antibody assay
* On a mycophenolate or azathioprine based immunosuppressive regimen
* > 6 months post-transplant

Exclusion Criteria:

* Pregnancy
* Contraindication to SARS-CoV-2 vaccination (severe allergic reactions or anaphylaxis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Change in anti-SARS-CoV-2 IgG titer to SARS-CoV-2 target proteins from baseline | 6 weeks after receipt of 3rd dose mRNA vaccine
Percentage of participants who achieve high-positive antibody titer | 6 weeks after receipt of 3rd dose mRNA vaccine

SECONDARY OUTCOMES:
Acute rejection | 1 week to 16 weeks after intervention
De Novo donor specific antibody (DSA) development | 4 week to 16 weeks after intervention
Change in donor-derived cell free DNA from baseline | 1 week to 16 weeks after intervention
Change in glomerular filtration rate (GFR) from baseline | 1 week to 16 weeks after intervention
Change in proteinuria from baseline | 1 week to 16 weeks after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan SF. Vaccination in kidney disease: what did we learn from COVID-19 pandemic. Curr Opin Nephrol Hypertens. 2023 Sep 1;32(5):412-417. doi: 10.1097/MNH.0000000000000901. Epub 2023 May 23. PMID 37382155